CLINICAL TRIAL: NCT05362708
Title: Neurophysiological Correlates of Dissociation Induced by Virtual Reality Hypnosis (VRH) in an Oncological Population
Brief Title: Neurophysiological Correlates of Dissociation Induced by Virtual Reality Hypnosis (VRH) in a Clinical Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Collaborators: Oncomfort (Industry); Biowin (Unknown)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, PhD, head of the Perception and Sensation Research Group - GIGA Consciousness, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: QuDDoS - Phase-II
Record Dates: First submitted 2022-04-13; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Cancer
Keywords: Virtual Reality; Hypnosis; Dissociation
MeSH Terms: conditions — Neoplasms; Dissociative Disorders | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Patients who are not interested will be considered as a control group.
Masking Description: Methodology of virtual reality hypnosis prevents masking participants and experimenter.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experimental group - VRH (Experimental): Patients will receive VRH during port-a-cath (Port) placement
  Interventions: Device: Clinical - Hypnosis with VR (VRH)
- Control Group (No Intervention): Patients who do not want to receive the VRH but who accept to answer the questionnaires will be considered as a control group.

INTERVENTIONS:
Device: Clinical - Hypnosis with VR (VRH) — The VRH intervention will use the Aqua video session developed by Oncomfort during a port-a-cath procedure.
  Arms: Experimental group - VRH

SUMMARY:
Hypnosis and virtual reality are potential tools for treating acute. Nevertheless, the neurophysiological correlates of such tools used together, i.e. 'virtual reality hypnosis' (VRH) (Patterson et al., 2004) remain mostly understudied. This study aims to improve our knowledge and understanding of the dissociation (i.e., a mental separation of components of behaviours that normally would be processed together) occurring during VRH. This is a clinical trial aiming at understanding if the VRH reduces pain during a port-a-cath intervention in oncological patients and if dissociation may explain the pain alteration.

DETAILED DESCRIPTION:
The study will be focused on oncological patients undergoing a port-a-cath placement procedure. Day-1 and Day-2 with a one-day follow-up Day-3:

I. Day-1: Oncological Population (Feasibility)

1. Recruitment and questionnaires on the day of the port-a-cath preparation consultation (DAY-1): i. A medical screening will be performed to assess eligibility, ii. Elkins Hypnotizability Scale. iii. State Trait Anxiety Inventory-trait (anxiety trait) iv. Dissociative Experience Scale. v. Tellegen Absorption Scale. vi. Questionnaire of Immersion Propensity.

II. Day-2:

1. Intervention day:

   i. Visual Analogy Scale:
   * Anxiety.
   * Pain. ii. 4-Electrodes EEG device from Oncomfort during port-a-cath (Port) placement procedure under Virtual Reality Hypnosis (VRH), combined standard monitoring (spO2, heart rate, etc.) iii. Adverse events will be recorded throughout the experiment iv. Visual Analogy Scale:
   * Dissociation.
   * Pain.
   * Anxiety
   * Absorption.
   * Arousal/wakefulness.
   * Automaticity v. Time Perception (open-ended question) vi. Presence questionnaire. vii. Satisfaction questionnaire.
2. Follow-up (DAY-3):

   i. A follow-up questionnaire using the Brief Pain Inventory (BPI) French version will be sent to the patient one week after the intervention to measure outcomes.

ELIGIBILITY:
Inclusion Criteria: Subject more than 18 years old

Exclusion Criteria:

1. Low auditory and/or visual acuity precludes the use of the device.
2. Head or face wounds precluding the use of the device.
3. Schizophrenia, dissociative disorder or any other psychiatric disorder.
4. Non-proficiency in French (Research language).
5. Patient under 18 years old.
6. Phobia of deep water.
7. Allergy to cutaneous electrodes.
8. Chronic pain and/or chronic analgesics consumption.
9. Medication affecting the autonomic nervous system.
10. Dizziness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Dissociation state | During the procedure
  Corresponds to a dissociation between the bodily sensations and the actual environment that one feels in a particular situation. will be assessed with a numerical rating scale (0= no dissociation; 10 = dissociation from environment).
Pain intensity | During the procedure
  The amount of pain one experiences in a particular situation. Will be assessed with a visual analogy scale, 0= no pain at all; 10= worst pain imaginable.

SECONDARY OUTCOMES:
Dissociation trait | During the procedure
  The amount of dissociation one experiences in one's daily life. Will be assessed with the Dissociative Experience Scale, the higher the score, the more one experiences dissociation in one's daily life.
Hypnotisability | During the procedure
  The susceptibility one has concerning hypnosis. Will be assessed with the Elkins Hypnotizability Scale. A score :
  0-3 : low hypnotizability 4-7: medium hypnotizability 8-11 : high hypnotizability 12 : very high hypnotizability
Absorption trait | During the procedure
  The tendency to become fully involved in a perceptual, imaginative or ideational experience. Will be assessed with the Tellegen Absorption Scale, the higher the score the higher the absorption in the daily life.
Anxiety trait | During the procedure
  Level of anxiety one experiences in one's daily life. Will be assessed with the State Trait Anxiety Invetory (STAI)-6 questionnaire. The higher the score, the higher the anxiety one feels in one's daily life.
Immersion propensity (trait) | During the procedure
  Immersion propensity is the amount of sensory input the virtual reality system creates. Will be assessed with the Immersion Propensity questionnaire. The higher the score, the more one is immersed in the virtual environments.
Anxiety state | During the procedure
  The amount of anxiety one experiences in a particular situation. Will be assessed with a visual analogy scale. a score = 0 means no anxiety at all, while a score = 10 means most anxiety ever felt.
Absorption state | During the procedure
  The amount of absorption one experiences in a particular situation. Will be assessed with a numerical rating scale, 0 = no absorption; 10 = fully absorption by the experience.
Automaticity | During the procedure
  A non-voluntary response related to the content of a communication that is intended to be a suggestion. Will be assessed with a numerical rating scale : 0= perfect control; 10 = passive witness.
Arousal/wakefulness | During the procedure
  The amount of arousal one experiences in a particular situation. Will be assessed with a visual analogy scale, 0=not aroused, awaken; 10 = completely aroused, awake.
Time perception | During the procedure
  Open-ended question about one's impression of the duration of the VHR and HYP sessions.
Cybersickness | During the procedure
  Assesses the sickness one might experience after the VRH. Will be assessed with the Cybersickness questionnaire. The higher the score, the more one has experience sickness during the VRH.
Presence | During the procedure
  Refers to the degree to which the subject experiences being in the virtual environment. Will be assessed with the presence questionnaire, the higher the score the higher one has the feeling of really being in the virtual environment.
Satisfaction of the participant | During the procedure
  Assesses the overall satisfaction one has had with the VRH and HYP session. Will be assessed by a self-made satisfaction questionnaire, the higher the score, the more one is satisfied with the experience.
Brief Pain Inventory | One week after the procedure
  The BPI measures the intensity of pain and interference of pain in the patient's life. The higher the scores the higher the intensity and interference.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey ANHAUDENHUYSE, PhD, Principal Investigator — CHU of Liège